CLINICAL TRIAL: NCT02670239
Title: Pharmacokinetics of Imipenem During Ex Vivo Lung Perfusion (EVLP)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Vito Fanelli MD, PhD, MD, PhD, University of Turin, Italy
Other Study IDs: CEI-178
Record Dates: First submitted 2016-01-22; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- EVLP group: All lungs from brain dead donors that were considered at high-risk for transplantation and underwent EVLP in the Turin lung transplantation program
  Interventions: Procedure: normothermic ex vivo lung perfusion

INTERVENTIONS:
Procedure: normothermic ex vivo lung perfusion

SUMMARY:
Ex vivo lung perfusion (EVLP) is an established strategy to evaluate and optimize high-risk donor lungs that would otherwise be rejected for transplantation mainly due to the presence of edema or infection. Extracorporeal circuits may negatively affects pharmacokinetic (PK) of several drugs including antibiotics, thus exposing patients to risk of therapeutic failure or drug toxicity. The investigators set out to examine the concentration of imipenem in lung perfusate and in lung biopsy during EVLP, and its clinical impact.

ELIGIBILITY:
Inclusion Criteria:

1. Best PaO2/FiO2 < 300 mmHg;
2. Pulmonary edema on chest X-Ray;
3. Poor inflation or deflation at visual inspection;
4. Need for blood transfusion of more than 10U;
5. Maastricht category III/IV

Exclusion Criteria:

1. Diagnosis of pneumonia;
2. severe mechanical injury;
3. gross gastric aspiration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: lungs from brain dead donors that were considered at high-risk for transplantation and underwent EVLP
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
imipenem concentration | change from baseline in imipenem concentration at 6 hours
  concentration of imipenem in lung perfusate and in lung biopsy during EVLP

SECONDARY OUTCOMES:
pathogens isolated from donors | 48 hours before lung procurement
pathogens isolated from recipients | 48 hours after lung transplantation
Clinical Pulmonary Infection Score | at 72 hours after lung transplantation
Primary graft dysfunction | at 72 hours after lung transplantation
Days of mechanical ventilation | at 28 days
Intensive Care Unit length of stay | at day 28

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Turin, Italy